CLINICAL TRIAL: NCT01418989
Title: An Open-label, Multi-center Study to Compare the Relative Bioavailability of Tocilizumab in Healthy Subjects Following Single Dose Subcutaneous (SC) Administration Via Disposable Auto-Injector (DAI) Device vs Pre-filled Glass Syringe (PFS)
Brief Title: A Study of Administration of RoActemra/Actemra (Tocilizumab) by Auto-injector Vs. Pre-filled Syringe in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP25539
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — tocilizumab; Syringes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra] auto-injector
- 2 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra] Syringe

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] Syringe — Single dose administration with pre-filled syringe
  Arms: 2
Drug: tocilizumab [RoActemra/Actemra] auto-injector — Single dose administration with auto-injector
  Arms: 1

SUMMARY:
This open-label, multi-center study will compare the bioavailability of RoActemra/Actemra (tocilizumab) administration by auto-injector versus pre-filled syringe in healthy volunteers. Healthy volunteers will receive a single dose of RoActemra/Actemra (tocilizumab). The anticipated time of study duration is 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, age 18 to 65 years inclusive
* Intact normal skin without potentially obscuring tattoos, pigmentation, lesion in the area for intended injection
* A body mass index (BMI) between 18 to 32 kg/m2 inclusive

Exclusion Criteria:

* Volunteers with any known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections
* A history of clinically significant gastrointestinal, renal, hepatic, cardiovascular, or allergic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of RoActemra/Actemra | 21 days
Peak plasma concentration of RoActemra/Actemra | 21 days

SECONDARY OUTCOMES:
Safety (Incidence of adverse events) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- France (2):
  - Montpellier
  - Rennes